CLINICAL TRIAL: NCT02527759
Title: Patient Self Monitoring to Evaluate 30 Day Post Discharge Heart Failure Outcomes
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0336
Record Dates: First submitted 2015-04-14; First posted 2015-08-19 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2016-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Survey

SUMMARY:
The purpose of this study is to examine the relative predictive ability of the derived monitoring instrument to determine post discharge instability and 30-day outcomes in patients discharged with HF. The primary hypothesis is that variables in the monitoring instrument, individually and combined, identify risk for 30-day outcomes. Clinical indicators of dyspnea, fatigue, orthopnea, dyspnea with exertion, daily weight, edema, heart rate, blood pressure, mental condition, medication adherence, and overall well-being will be reported by participants on a daily basis and considered indicators for 30-day outcomes of stability, re-hospitalization, or mortality.

ELIGIBILITY:
Inclusion Criteria:

1. > 65 years of age
2. male and female patients admitted to the hospital with the primary diagnosis of HF with hospitalization > 24 hours
3. able to read and write in English
4. discharged to home environment

Exclusion Criteria:

1. a cardiac transplant candidate
2. experienced an acute coronary event within the previous 30 days of index hospitalization
3. experienced percutaneous coronary intervention or coronary artery bypass grafting within the previous 30 days of index hospitalization
4. end stage renal disease/hemodialysis
5. have a left ventricular assist device
6. > 400 lbs
7. unable to stand for 90 seconds independently

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events of rehospitalization and/or mortality. | 30 days
  Trial a novel 30-day post-discharge monitoring instrument after hospitalization for heart to evaluate patient status based on patient self-monitoring.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medstar, Washington Hospital Center, Washington D.C., District of Columbia
  - Medstar, Georgetown University Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.